CLINICAL TRIAL: NCT03948347
Title: Liraglutide in Acute Minor Ischemic Stroke or High-risk Transient Ischemic Attack Patients With Type 2 Diabetes Mellitus: A Prospective, Multicenter, Randomized, Blank-controlled，Blinded End-point Study.
Brief Title: Liraglutide in Acute Minor Ischemic Stroke or High-risk Transient Ischemic Attack Patients With Type 2 Diabetes Mellitus
Acronym: LAMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Jinan University (Other)
Responsible Party: Principal Investigator, Anding Xu, Dean of the First Affiliated Hospital of Jinan University, First Affiliated Hospital of Jinan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LAMP20190508
Record Dates: First submitted 2019-05-10; First posted 2019-05-13 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack; Type 2 Diabetes Mellitus
Keywords: ischemic stroke; transient ischemic attack; glucagon-like peptide-1; type 2 diabetes mellitus
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active (Active Comparator): Active patients will receive liraglutide injections
  Interventions: Drug: Liraglutide
- standard care/no intervention (No Intervention): standard care for stroke as per hospital protocol

INTERVENTIONS:
Drug: Liraglutide — The treatment arm will receive the starting dose of liraglutide of 0.6 mg/d subcutaneously once daily, and the dose will be increased to 1.8 mg/d in two weeks, and then continue to administrate this dose for 90 days.
  Other Names: Victoza
  Arms: active

SUMMARY:
The purpose of this study is to assess the safety and efficacy of glucagon-like peptide-1 (GLP-1) analogue liraglutide in the treatment of acute minor stroke (National Institute of Health stroke scale, NIHSS ≤ 3) or high-risk transient ischemic attack (TIA) (ABCD2 score ≥ 4 ) patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
The treatment arm will receive the starting dose of liraglutide of 0.6mg/d subcutaneously once daily, and the dose will be increased to 1.8mg/d in two weeks, and then continue to administrate this dose for 90 days. The control arm will not use liraglutide. Other types of GLP-1 analogues or degraded by dipeptidyl peptidase-IV (DPP-IV) inhibitors will be prohibited. Study visits will be performed at day 7, day 30±3 and at 90±7 day.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (male or female ≥ 50 years);
* Acute ischemic stroke patients (NIHSS ≤ 3 at the time of randomization) with type 2 diabetes mellitus within 24 hours of symptoms onset;
* High-risk TIA patients (ABCD2 score ≥ 4 at the time of randomization) with type 2 diabetes mellitus within 24 hours of onset;
* First stroke, or prior stroke without sequel (mRS score ≤ 1) and does not affect the NIHSS score;
* Informed consent signed.

Exclusion Criteria:

* Diagnosis of hemorrhage brain disease on baseline head CT;
* Iatrogenic and cardiogenic stroke;
* Patients receiving thrombolysis or endovascular treatment;
* Use of a GLP-1 analogue or any dipeptidyl peptidase-IV (DPP-IV) inhibitor within the 3 months prior to screening;
* Family or personal history of multiple endocrine neoplasia type 2 (MEN2) or familial medullary thyroid carcinoma (FMTC);
* Patients with pancreatitis or previous history of pancreatitis, inflammatory bowel disease and gastroparesis;
* Pregnant, lactating women,or patients who are likely to have a pregnancy and plan to have one;
* Allergic to liraglutide or excipients;
* Congestive heart failure (NYHA class III-IV);
* Severe liver and kidney dysfunction (AST/ALT is 3 times higher than the normal upper limit, serum creatinine is 3 times higher than the normal upper limit);
* Patients with malignant tumors who are expected to have a survival period of less than three months;
* Participated in other clinical trials of drugs within 3 months;
* Researchers believe that patients who are not suitable for this clinical study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1708 (Estimated)
Dates: Start 2019-06-25 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with the 90-day new stroke events (ischemic or hemorrhagic) | 90 days
  Definition of ischemic stroke: An episode of neurological dysfunction caused by focal cerebral, spinal, or retinal infarction. Either of the following is considered to be an ischemic stroke: a new focal neurologic deficit lasting for less than 24 hours and not attributable to a nonischemic cause but accompanied by neuroimaging evidence of new brain infarction; sudden onset of a new focal neurologic deficit, with clinical or imaging evidence of infarction lasting 24 hours or more and not attributable to a nonischemic cause.
  Definition of hemorrhagic stroke: Rapidly developing clinical signs of neurological dysfunction attributable to a focal collection of blood within the brain parenchyma, ventricular system or subarachnoid space that is not caused by trauma.

SECONDARY OUTCOMES:
Percentage of patients with the 90-day new clinical vascular events (ischemic stroke/hemorrhagic stroke/TIA/myocardial infarction/vascular death) | 90 days
  Transient ischemic attack was defined as transient neurological deficits caused by focal brain or retinal ischemia, the clinical symptoms are generally no more than 1 hour, and the longest duration is less than 24 hours, and there is no evidence of a responsible lesion.
  The clinical definition of myocardial infarction denotes the presence of acute myocardial injury detected by abnormal cardiac biomarkers in the setting of evidence of acute myocardial ischemia.
  Vascular death was defined as death due to stroke (ischemic or hemorrhagic), systemic hemorrhage, myocardial infarction, congestive heart failure, pulmonary embolism, sudden death, or arrhythmia.
Percentage of patients with the 90-day Modified Rankin Scale (mRS) ≤ 2 | 90 days
  The modified Rankin scale is used to measure the recovery of neurological function in patients after stroke. The following questionnaire will be used to determine the mRs score:
  The modified Rankin scale is used to measure the recovery of neurological function in patients after stroke. The following questionnaire will be used to determine the mRs score:
  0- No symptoms at all.
  1. No significant disability despite symptoms; able to carry out all usual duties and activities.
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance.
  3. Moderate disability; requiring some help, but able to walk without assistance.
  4. Moderately severe disability, unable to walk without assistance and unable to attend to own bodily needs without assistance.
  5. Severe disability, bedridden, incontinent and require constant nursing care and attention.
  6. Dead.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhu H, Yang B, Lu L, Li Y, Sui R, Liu K, Tan S, Wang L, Qiu J, Zhong J, Wei T, Bei Y, Huang J, Zhang S, Ji Y, Wu W, Li Y, Huang Y, Chen Y, Huang X, Zeng G, Zhang Y, Huang L, Li H, Wang X, Wang Y, Xu A; LAMP Investigators. Liraglutide in Acute Minor Ischemic Stroke or High-Risk Transient Ischemic Attack With Type 2 Diabetes: The LAMP Randomized Clinical Trial. JAMA Intern Med. 2026 Jan 1;186(1):46-54. doi: 10.1001/jamainternmed.2025.5684. PMID 41182740